CLINICAL TRIAL: NCT06461689
Title: Comparison of Changes in Tumor Burden (Toral Tumor Volume [TMTV] and Total Lesion Activity [TLA]) in 68Ga-PSMA-11 PET/CT and 177Lu-PSMA SPECT/CT in the Monitoring of Metastatic Castration-resistant Prostate Cancer Treated With 177Lutetium-PSMA-617
Brief Title: Comparison of Changes in Tumor Burden in 68Ga-PSMA-11 PET/CT and 177Lu-PSMA SPECT/CT in Metastatic Castration-resistant Prostate Cancer
Acronym: PROLUT
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BOURSIER Caroline, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2024PI106
Record Dates: First submitted 2024-06-05; First posted 2024-06-17 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer Metastatic
Keywords: prostate cancer; theragnostic
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pluvicto

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient treated as part of mCPRC: All patients treated with 177Lu-PSMA had post-therapy 68Ga-PSMA PET and 177Lu-PSMA-617 SPECT/CT.
  Interventions: Drug: 177Lu-PSMA-617

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — All patients treated with 177Lu-PSMA had a post-therapy 68Ga-PSMA PET scan and a post-therapy 177Lu-PSMA-617 SPECT/CT scan. These scans are available in the CHRU PACS, and patients are informed that their data may be used for research purposes, via posters in the nuclear medicine department or via the welcome booklet,

SUMMARY:
To demonstrate the prognostic value of using post-therapy 177Lu-PSMA SPECT/CT versus 68Ga-PSMA-11 PET/CT in mCPRC patients progressing despite chemotherapy and treated with 177Lu-PSMA.

DETAILED DESCRIPTION:
Since few years, therapy by 177Lu-PSMA in nancy hospital began. A lot's of datas were collected. Prostate cancer is the number one killer in france and this is very important to find a diagnostic tool.

The hypothesis of this study is to demonstrate the prognostic value of using post-therapy 177Lu-PSMA SPECT/CT versus 68Ga-PSMA-11 PET/CT in mCPRC patients progressing despite chemotherapy and treated with 177Lu-PSMA.

ELIGIBILITY:
Inclusion Criteria:

* patient who received a dose of 177lu-PSMA
* patient who had imaging by 68Ga-PSMA
* patient treated in Nancy hospital for its cancer prostate

Exclusion Criteria:

* no social security
* no acceptation to participating in retrospective study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients treated with 177Lu-PSMA had post-therapy 68Ga-PSMA PET and 177Lu-PSMA-617 SPECT/CT.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Measurement of TMTV (total metabolic tumor volume) | 12 months
  Measurement of TMTV (total metabolic tumor volume) on 68Ga-PSMA-11 PET/CT (pre-treatment, after 4th treatment and after 6th treatment) and on SPECT/CT (after each treatment).
Measurement of TLA (total lesion activity) | 12 months
  Measurement of TLA (total lesion activity) on 68Ga-PSMA-11 PET/CT (pre-treatment, after 4th treatment and after 6th treatment) and on SPECT/CT (after each treatment).

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de NANCY, Vandœuvre-lès-Nancy, France